CLINICAL TRIAL: NCT03657173
Title: Ultrasound Image Quality of the Brachial Plexus at the Interscalene Space Before and After Shoulder Arthroscopy: a Prospective Cohort Study
Brief Title: Ultrasound Image Quality of the Brachial Plexus at the Interscalene Space Before and After Shoulder Arthroscopy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bridget P. Pulos, Principal Investigator, Mayo Clinic
Other Study IDs: 18-004131
Record Dates: First submitted 2018-08-27; First posted 2018-09-04 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ultrasound guided interscalene nerve blockade with local anesthesia is a standard regional anesthetic technique for providing postoperative analgesia during shoulder arthroscopy and wide variety of shoulder procedures. There is a paucity of data regarding the effects of shoulder arthroscopy on ultrasound image quality, including the effects of muscle mobilization and the use of large volume irrigation and subsequent tissue absorption, though increased neck circumference and airway edema are known complications of arthroscopic shoulder procedures.

The objective of the study is to determine if there is a difference in ultrasound image quality of the interscalene block anatomy, by Likert scale, pre- versus post-operatively in a cohort of patients undergoing shoulder arthroscopy who routinely receive blockade of the brachial plexus for postoperative analgesia. Further, if there are differences in imaging quality, correlations with surgical and patient factors will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing shoulder procedures involving arthroscopy
* Subject has consented to interscalene blockade for postoperative analgesia

Exclusion Criteria:

* Patient refusal
* Contraindications to interscalene blockade, including significant pulmonary insufficiency, hemi-diaphragmatic paralysis, brachial plexus or degenerative neuropathy
* Allergy to proposed local anesthetic medication\
* Severe cervical spine disease.
* BMI >40 kg/m2
* Neck Circumference > 50cm
* Failed preoperative interscalene blockade
* Patients known to be currently pregnant or actively breastfeeding
* Patients where English is a language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years of age) undergoing shoulder procedures involving arthroscopy who have consented to interscalene blockade for postoperative analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Likert Scale | 2-3 months
  Ultrasound media will be scored using a Likert scale (from 1-5 based on quality of imaging) individually for pre-operative and post-operative scanning for each enrolled patient

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Panchamia JK, Jagannathan R, Pulos BP, Amundson AW, Sanchez-Sotelo J, Martin DP, Smith HM. The effects of shoulder arthroscopy on ultrasound image quality of the interscalene brachial plexus: a pre-procedure vs post-procedure comparative study. BMC Anesthesiol. 2021 Jul 9;21(1):187. doi: 10.1186/s12871-021-01409-3. PMID 34243720